CLINICAL TRIAL: NCT02713139
Title: Phase III, Multicenter, Randomized, Parallel, Open Label, Controlled and Comparative Study to Evaluate the Efficacy and Safety of the Association of Clotrimazole 200mg and Metronidazole 0,75% (Colpistatin 5DT®) Compared to Gynecological Flagyl®(Metronidazole 100mg/g) and the Vaginal Cream Gino-Canesten® 3 (Clotrimazole 20mg/g) in the Syndromic Treatment of the Vaginal Discharge From Different Etiologies.
Brief Title: Efficacy and Safety of the Association of Clotrimazole and Metronidazole in the Treatment of Vaginal Discharge From Different Etiologies.
Acronym: Frauen
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to budget limitations, the company decided to withdraw this study.
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CLP-03(05/12)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Sexual Active Women; Vaginal Discharge
Keywords: vaginal; discharge; women
MeSH Terms: conditions — Vaginal Discharge | interventions — Clotrimazole; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Colpistatin 5DT (Experimental)
  Interventions: Drug: Clotrimazole + Metronidazole
- Gynecological Flagyl (Active Comparator)
  Interventions: Drug: Metronidazole
- Gino-Canesten 3 (Active Comparator)
  Interventions: Drug: Clotrimazole

INTERVENTIONS:
Drug: Clotrimazole + Metronidazole — Vaginal cream with Clotrimazole 200mg and Metronidazole 0,75%. Apply once per day, before bedtime, for 5 (five) days.
  Arms: Colpistatin 5DT
Drug: Metronidazole — Vaginal gel with Metronifdazole 100mg/g. Apply once per day, before bedtime, for 10(ten) days.
  Arms: Gynecological Flagyl
Drug: Clotrimazole — Vaginal cream with Clotrimazole 20mg/g. Apply once per day, before bedtime, for 3 (three) days.
  Arms: Gino-Canesten 3

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the association clotrimazole 200mg and metronidazole 0,75%(Clopistatin 5DT®) and whether it is superior when compared with metronidazole 100mg/g (gynecologic Flagyl®) and clotrimazole 20mg/g (Gino-Canesten® 3) in the syndromic treatment of vaginal discharge from different etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that have already started sexual activity;
* Subjects with complaints of vaginal discharge and had not received treatment in the 30 days before the enrollment visit;
* Subjects in the premenopausal period must be under usage of acceptable contraceptive methods(oral contraceptive, injectable contraceptives, IUD, hormonal implant, hormone transdermal adhesive, tubal ligation) or are surgically sterile (bilateral oophorectomy or hysterectomy); or accept to utilize a barrier contraceptive provided by the sponsor during the period of the study;
* Subjects with the capacity to comprehend and understand her participation in this clinical trial, manifested through informed consent form, even if with the help of another person (Legal representative).

Exclusion Criteria:

* Subjects with chronic diseases (diabetes mellitus, neoplasia, renal failure, tuberculosis) or any clinical and/or laboratory find (anamnesis, physical exam and/or laboratory tests) that is interpreted, in the investigator's opinion, as a risk to the subject's participation in the clinical trial;
* Menopausal women;
* Known hyper-sensibility to any of the products' components;
* Pregnant or lactating women;
* Subjects with active genital ulcer and/or with Genital herpes diagnosis;
* Diagnosis or suspicion of Inflammatory pelvic disease;
* Diagnosis of Vulvar condyloma acuminata;
* Subjects under the usage of systemic corticosteroids for a period superior than 2 (two) months or under the usage of chemotherapeutics;
* Transplanted subjects;
* Subjects with history of active autoimmune diseases or with immune suppression;
* Subjects under the usage of medication or therapy described on the protocol item "Prohibited Treatments";
* Subjects that have participated on a clinical trial in the last 12 months (Conselho Nacional de Saúde - Resolução 251, de 7 de agosto de 1997, item III, sub-item J), unless the subject can have a direct benefit, in the investigator opinion;
* Subject that have a kinship or bond with any employees of Sponsor or Research center;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Ceasing of the symptoms of vaginal discharge after 3(three) days of the end of the treatment | From baseline to 3 days after the end of the treatment
  Examination of the breasts and internal and external examination of the female genital organ.

SECONDARY OUTCOMES:
Registry of Adverse Effects occurrence throughout the study | From baseline to 30 days after the end of the treatment
  Evaluation of Clinical and Physical examination and the measure of vital signs; Evaluation of Adverse effects; Evaluation of Laboratory exams; And evaluation of urine beta-hcg test.
Vaginal microflora reconstitution through microbiological evaluation of vaginal material | From baseline to 30 days after treatment's end
  Evaluation of the collected vaginal material with the microbiological tests(Whiff, Gram, Affirm VPIII) and PCR.
Symptomatology recurrence and/or vaginal microflora alteration 30 days after the treatment's end | From baseline to 30 days after treatment's end
  Examination of the breasts and internal and external examination of the female genital organ.
  Evaluation of the collected vaginal material with the microbiological tests(Whiff, Gram, Affirm VPIII) and PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo A. Junior, MD, Principal Investigator — Scentryphar Pesquisa Clínica Ltda